CLINICAL TRIAL: NCT03696199
Title: A Prospective, Randomized Trial Evaluating Regional Anesthesia, Long-Acting Local Anesthesia, and Traditional Care for Pain Control of Operatively Treated Ankle Fractures
Brief Title: Randomized Controlled Trial for Ankle Fracture Pain Control
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Eric Francis Swart, Principal Investigator, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20223040
Record Dates: First submitted 2018-09-24; First posted 2018-10-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Traditional Pain Control Care (No Intervention): Standard of care post-operative pain control with oral narcotics
- Regional Anesthesia (Experimental): Single injection perioperative peripheral nerve block + followed by administration of oral narcotics on a need-based system
  Interventions: Drug: Regional Anesthesia
- Long-Acting Local Anesthesia (Experimental): Subcutaneous local cocktail injection + followed by administration of oral narcotics on a need-based system
  Interventions: Drug: Long-Acting Local Anesthesia

INTERVENTIONS:
Drug: Long-Acting Local Anesthesia — The cocktail consists of:
  * 0.5% Ropivicaine, 24.6 mL
  * Clonidine 100 mcg/mL, 0.4mL
  * Epinephrine 1mg/mL, 0.5mL
  * Saline to total volume of 50 mL (24.5mL of saline)
  The total amount of solution prepared is 50mL, but typically 30mL is used based on the size of the incision. The total volume administered will be recorded.
  Other Names: Local Cocktail
  Arms: Long-Acting Local Anesthesia
Drug: Regional Anesthesia — 0.5% ropivicaine - 30mL each sciatic and femoral/saphenous nerve, ultrasound guided
  Other Names: Ropivicaine
  Arms: Regional Anesthesia

SUMMARY:
This project is a multicenter, three armed, prospective randomized control trial studying the effectiveness of a long-acting local anesthetic "cocktail" in patients undergoing operative fixation of ankle fractures.

DETAILED DESCRIPTION:
This study is a multicenter, three armed, prospective randomized control trial studying the effect of a long-acting local anesthetic "cocktail" in patients undergoing operative fixation of ankle fractures.

Primary Hypothesis Driven Aims:

1. Determine the effectiveness of a local anesthesia "cocktail" compared to regional block or standard of care in controlling pain in operatively treated ankle fractures. Nearly one out of ten fractures treated by both orthopaedic traumatologists and general orthopaedic surgeons taking call are ankle fractures. As such, effective pain control in this group of patients represents an opportunity to make a large impact, especially in the context of the current opioid epidemic. Improved pain control can help improve patient satisfaction, outcomes, decrease length of stay, cost of care, and complications associated with traditional narcotic use.

   * Hypothesis 1A: Patients receiving the intraoperative cocktail will have improved post-operative pain control compared to those receiving a peri-operative nerve block or standard of care.
   * Hypothesis 1B: Patients receiving the intraoperative cocktail or peri-operative nerve block will have improved post-operative pain control when compared to standard of care.
   * Null Hypothesis 1: There will be no difference in post-operative pain control between all treatment arms.
2. Determine the economic impact of cocktail and regional blocks in ankle fractures. A common concern with the use of regional blocks is the cost of the additional procedure, along with logistic delays which are associated with coordinating a separate procedure. This study would provide valuable data about the additional costs associated with regional blocks and with cocktail administration which could help aid in making economically conscious treatment decisions.

   * Hypothesis 2: Local cocktail administration will have significantly lower costs than regional block, and not be significantly more expensive than standard of care.
   * Null Hypothesis 2: There is no difference in cost between the modalities.

Secondary Aim:

Demonstrate the use of long-acting local anesthetic as a viable pain management strategy in fracture surgery. Although long-acting local anesthetics have an established track record in arthroplasty, there is a paucity of evidence guiding their use in fractures. Small case series in trauma and foot/ankle patients have been encouraging, but a rigorously conducted, prospective trial in a relatively homogeneous group could generate pilot data to validate the use of long acting local anesthetics in fracture surgery. This knowledge may be translatable to other extremity injuries as well, having a greater impact than the scope of the proposed trial.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a bimalleolar ankle fracture (OTA/AO type 44 A2, B2, C1, and C2 fracture) with surgery indicated and an approach with medial and lateral incisions planned Syndesmotic injuries will be included, due to the practical difficulty of reliably determining the presence of a syndesmotic injury preoperatively Trimalleolar ankle fractures where fixation of the posterior malleolus is not planned will also be included
* Isolated Injury

Exclusion Criteria:

* Unifocal malleolar fractures
* Bimalleolar fractures where fixation of only one malleolus is planned
* Posterior malleolus fractures requiring fixation
* Patients ineligible for a peripheral nerve block (e.g. concern for compartment syndrome)
* Open injury
* Patients treated with external fixation
* Neurologic condition that would confound results (e.g. peripheral neuropathy)
* Inability to consent
* Chronic opioid use
* History of opiate abuse
* Polytrauma as defined as additional boney injury, visceral injury or moderate soft tissue injury (requiring suture repair or other invasive procedure)
* Prisoners (unlikely to be accessible for follow-up)
* Pregnant patients
* Non-English-speaking subjects (post-operative data collection procedure involves conversations via phone calls. As we do not have access to translators for this research project, we will work exclusively with English-speaking subjects).
* Subjects unable to take the standard post-operative pain regimen that consists of gabapentin, oxycodone, acetaminophen, and ibuprofen.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Oral Narcotics / Morphine Milligram Equivalents (MME) given | 72 postoperative hours
  The medical record (EPIC) will be used to determine the total morphine equivalents given to the patient post-surgery, including recovery unit administration of narcotics in the immediate post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swart, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

REFERENCES:
- [Background] Barrington JW, Olugbode O, Lovald S, Ong K, Watson H, Emerson RH Jr. Liposomal Bupivacaine: A Comparative Study of More Than 1000 Total Joint Arthroplasty Cases. Orthop Clin North Am. 2015 Oct;46(4):469-77. doi: 10.1016/j.ocl.2015.06.003. Epub 2015 Aug 6. PMID 26410636
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Ng FY, Ng JK, Chiu KY, Yan CH, Chan CW. Multimodal periarticular injection vs continuous femoral nerve block after total knee arthroplasty: a prospective, crossover, randomized clinical trial. J Arthroplasty. 2012 Jun;27(6):1234-8. doi: 10.1016/j.arth.2011.12.021. Epub 2012 Feb 8. PMID 22325963
- [Background] Lonner J. Role of liposomal bupivacaine in pain management after total joint arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):37-41. doi: 10.3113/jsoa.2014.0037. PMID 24641895
- [Background] Hutchinson HL. Local infiltration of liposome bupivacaine in orthopedic trauma patients: case-based reviews. Am J Orthop (Belle Mead NJ). 2014 Oct;43(10 Suppl):S13-6. PMID 25303455
- [Background] Herbst SA. Local infiltration of liposome bupivacaine in foot and ankle surgery: case-based reviews. Am J Orthop (Belle Mead NJ). 2014 Oct;43(10 Suppl):S10-2. PMID 25303454
- [Background] Stein BE, Srikumaran U, Tan EW, Freehill MT, Wilckens JH. Lower-extremity peripheral nerve blocks in the perioperative pain management of orthopaedic patients: AAOS exhibit selection. J Bone Joint Surg Am. 2012 Nov 21;94(22):e167. doi: 10.2106/JBJS.K.01706. PMID 23172334
- [Background] Wang J, Liu GT, Mayo HG, Joshi GP. Pain Management for Elective Foot and Ankle Surgery: A Systematic Review of Randomized Controlled Trials. J Foot Ankle Surg. 2015 Jul-Aug;54(4):625-35. doi: 10.1053/j.jfas.2014.05.003. Epub 2014 Jun 18. PMID 24954920
- [Background] Compton P, Athanasos P. Chronic pain, substance abuse and addiction. Nurs Clin North Am. 2003 Sep;38(3):525-37. doi: 10.1016/s0029-6465(02)00100-7. PMID 14567207
- [Background] De Maeyer J, Vanderplasschen W, Broekaert E. Quality of life among opiate-dependent individuals: A review of the literature. Int J Drug Policy. 2010 Sep;21(5):364-80. doi: 10.1016/j.drugpo.2010.01.010. Epub 2010 Feb 20. PMID 20172706
- [Background] Morrone LA, Scuteri D, Rombola L, Mizoguchi H, Bagetta G. Opioids Resistance in Chronic Pain Management. Curr Neuropharmacol. 2017 Apr;15(3):444-456. doi: 10.2174/1570159X14666161101092822. PMID 28503117
- [Background] Holman JE, Stoddard GJ, Higgins TF. Rates of prescription opiate use before and after injury in patients with orthopaedic trauma and the risk factors for prolonged opiate use. J Bone Joint Surg Am. 2013 Jun 19;95(12):1075-80. doi: 10.2106/JBJS.L.00619. PMID 23783203
- [Background] Manchikanti L. National drug control policy and prescription drug abuse: facts and fallacies. Pain Physician. 2007 May;10(3):399-424. PMID 17525776
- [Background] Elkassabany N, Cai LF, Mehta S, Ahn J, Pieczynski L, Polomano RC, Picon S, Hogg R, Liu J. Does Regional Anesthesia Improve the Quality of Postoperative Pain Management and the Quality of Recovery in Patients Undergoing Operative Repair of Tibia and Ankle Fractures? J Orthop Trauma. 2015 Sep;29(9):404-9. doi: 10.1097/BOT.0000000000000344. PMID 25882965
- [Background] Cometa MA, Esch AT, Boezaart AP. Did continuous femoral and sciatic nerve block obscure the diagnosis or delay the treatment of acute lower leg compartment syndrome? A case report. Pain Med. 2011 May;12(5):823-8. doi: 10.1111/j.1526-4637.2011.01109.x. PMID 21564511
- [Background] Mar GJ, Barrington MJ, McGuirk BR. Acute compartment syndrome of the lower limb and the effect of postoperative analgesia on diagnosis. Br J Anaesth. 2009 Jan;102(1):3-11. doi: 10.1093/bja/aen330. Epub 2008 Nov 19. PMID 19022795
- [Background] Goldstein RY, Montero N, Jain SK, Egol KA, Tejwani NC. Efficacy of popliteal block in postoperative pain control after ankle fracture fixation: a prospective randomized study. J Orthop Trauma. 2012 Oct;26(10):557-61. doi: 10.1097/BOT.0b013e3182638b25. PMID 22732860
- [Background] Ding DY, Manoli A 3rd, Galos DK, Jain S, Tejwani NC. Continuous Popliteal Sciatic Nerve Block Versus Single Injection Nerve Block for Ankle Fracture Surgery: A Prospective Randomized Comparative Trial. J Orthop Trauma. 2015 Sep;29(9):393-8. doi: 10.1097/BOT.0000000000000374. PMID 26165259
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Schroer WC, Diesfeld PG, LeMarr AR, Morton DJ, Reedy ME. Does Extended-Release Liposomal Bupivacaine Better Control Pain Than Bupivacaine After Total Knee Arthroplasty (TKA)? A Prospective, Randomized Clinical Trial. J Arthroplasty. 2015 Sep;30(9 Suppl):64-7. doi: 10.1016/j.arth.2015.01.059. Epub 2015 Jun 3. PMID 26117072
- [Background] Bagsby DT, Ireland PH, Meneghini RM. Liposomal bupivacaine versus traditional periarticular injection for pain control after total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1687-90. doi: 10.1016/j.arth.2014.03.034. Epub 2014 Apr 4. PMID 24793570
- [Background] Joshi GP, Cushner FD, Barrington JW, Lombardi AV Jr, Long WJ, Springer BD, Stulberg BN. Techniques for periarticular infiltration with liposomal bupivacaine for the management of pain after hip and knee arthroplasty: a consensus recommendation. J Surg Orthop Adv. 2015 Spring;24(1):27-35. PMID 25830260
- [Background] Kelley TC, Adams MJ, Mulliken BD, Dalury DF. Efficacy of multimodal perioperative analgesia protocol with periarticular medication injection in total knee arthroplasty: a randomized, double-blinded study. J Arthroplasty. 2013 Sep;28(8):1274-7. doi: 10.1016/j.arth.2013.03.008. Epub 2013 Apr 20. PMID 23608085
- [Background] Zhao X, Qin J, Tan Y, Mohanan R, Hu D, Chen L. Efficacy of steroid addition to multimodal cocktail periarticular injection in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2015 May 22;10:75. doi: 10.1186/s13018-015-0214-8. PMID 25994175
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Myles PS, Reeves MD, Anderson H, Weeks AM. Measurement of quality of recovery in 5672 patients after anaesthesia and surgery. Anaesth Intensive Care. 2000 Jun;28(3):276-80. doi: 10.1177/0310057X0002800304. PMID 10853209

DOCUMENTS (1):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03696199/Prot_000.pdf